CLINICAL TRIAL: NCT02677597
Title: An Open, Multicenter, Randomized Phase III Clinical Study on Cisplatin Combined With S-1 or Paclitaxel as First-line Treatment for Metastatic Esophageal Squamous Cell Carcinoma
Brief Title: Cisplatin Combined With S-1 or Paclitaxel as First-line Treatment for Metastatic Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Chang Jian Hua, Chief Physician, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CISPEC study
Record Dates: First submitted 2016-02-05; First posted 2016-02-09 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — S 1 (combination); Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cisplatin Combined With S-1 (Experimental): Cisplatin 75mg/m2 ivgtt d1 S-1 BSA<1.5 50mg bid，BSA≥1.5 60mg bid po d1-14
  Interventions: Drug: Cisplatin Combined With S-1
- Cisplatin Combined With Paclitaxel (Experimental): Cisplatin 75mg/m2 ivgtt d1 Paclitaxel 175mg/m2 d1 ivgtt 3h
  Interventions: Drug: Cisplatin Combined With Paclitaxel

INTERVENTIONS:
Drug: Cisplatin Combined With S-1
  Arms: Cisplatin Combined With S-1
Drug: Cisplatin Combined With Paclitaxel
  Arms: Cisplatin Combined With Paclitaxel

SUMMARY:
Cisplatin Combined With S-1 or Paclitaxel as First-line Treatment for Metastatic Esophageal Squamous Cell Carcinoma

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven primary thoracic esophageal squamous cell carcinoma
* Not suitable for surgery or radio or chemical therapy
* Presence of at least one index lesion measurable by CT scan or MRI radiation therapy ended at least 4 weeks, but part of the radiation does not as a measurable lesions
* 18~70 years
* PS:0-1
* Life expectancy of ≥ 3 months
* WBC≥3.5×109/L,ANC≥1.5×109/L, PLT≥100×109/L, Hb≥100g/L
* TB ≤ 1.5UNL, ALT/AST ≤ 2.5×UNL
* Scr≥60 mL/min
* Normal electrocardiogram (ecg)
* Can normal oral drugs
* Signed written informed consent

Exclusion Criteria:

* Breast-feeding or pregnant women, no effective contraception if risk of conception exists
* Chronic diarrhea, enteritis, intestine obstruction which are not under control
* Esophageal obstruction cannot eat liquid completely, esophagus have deep ulcer perforation or hematemesis; Esophageal cancer common complications such as anastomotic leakage, serious lung complications, etc.
* A second primary tumor (except skin basal cell carcinoma)
* The original serious heart disease, including: higher risk of congestive heart failure, unable to control arrhythmia, unstable angina, myocardial infarction, severe valvular heart disease, and resistant hypertension
* With uncontrol nerve, mental illness or mental disorders, compliance is poor, can't cooperate with accounts and response to treatment; Primary brain tumors or - CNS metastases illness did not get a control, has obvious cranial hypertension or nerve mental symptoms
* With bleeding tendency
* Has inherited bleeding evidence of physical or blood coagulation disorder
* With clear chemotherapy drug allergy
* Other researchers believe that patients should not participate in this testing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
PFS | Since the date of random to disease progression or any cause of death，the average time is 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes